CLINICAL TRIAL: NCT05781022
Title: Endoscopic Management Of Iatrogenic Esophageal Perforation After Laparoscopic Upper Gastrointestinal Surgery : A Randomized Controlled Trial.
Brief Title: Endoscopic Management Of Iatrogenic Esophageal Perforation After Laparoscopic Upper Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: esophageal injury
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Iatrogenic Esophageal Perforation
Keywords: stent, endoscopy , esophagus , iatrogenic injury

STUDY DESIGN:
Intervention Model Description: The investigators included all patients who were presented to General Surgery Department with Iatrogenic Esophageal Perforation after Laparoscopic Upper Gastrointestinal Surgery at Zagazig University hospital between (December 2020 to August 2023).Patients will be divided into 2 groups in accordance type of preoperative
  Therapy :
  Group 1: "Endoscopic Group, EG" included 42 patients. Group 2: "Surgical Group , SG" included 42 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) endoscopic group (Active Comparator): For patients in EG, we began with assessment of the site & size of perforation . In this study, In this study, we used a fully covered stent (Mega stent, Taewoong Medical Industries, Gyeonggi-do, South Korea) ultra large and long (length: 24 cm, diameter: 36 mm) stent. We did not experience any complication with Mega stent, particularly migration, thanks to the design of Mega stent that fits well for the post-sleeve anatomy with reduction of migration.
  Concurrently, the interventional radiology team subcutaneously drained the intraperitoneal free fluid using 2 intra-peritoneal tubes that were placed under US guidance in the sub-hepatic region and in the pelvis
  Interventions: Procedure: endoscopic repair of iatrogenic esophageal perforation
- group (2) surgical group (No Intervention): surgical repair of perforation after adequate drainage

INTERVENTIONS:
Procedure: endoscopic repair of iatrogenic esophageal perforation — For patients in EG, we began with assessment of the site & size of perforation . In this study, In this study, we used a fully covered stent (Mega stent, Taewoong Medical Industries, Gyeonggi-do, South Korea) ultra large and long (length: 24 cm, diameter: 36 mm) stent. We did not experience any complication with Mega stent, particularly migration, thanks to the design of Mega stent that fits well for the post-sleeve anatomy with reduction of migration.
  Concurrently, the interventional radiology team subcutaneously drained the intraperitoneal free fluid using 2 intra-peritoneal tubes that were placed under US guidance in the sub-hepatic region and in the pelvis
  Arms: group (1) endoscopic group

SUMMARY:
The investigators included all patients who were presented to General Surgery Department with Iatrogenic Esophageal Perforation after Laparoscopic Upper Gastrointestinal Surgery at Zagazig University hospital between (December 2020 to August 2023).The sample size was calculated by using open Epi program depending on the following data ; confidence interval 95% , power of the test 80% , ratio of unexposed/ exposed 1 , the success rate of surgical repair versus endoscopic repair was 98 % versus 75% respectively. Odd ratio 16 , and risk ratio 1.3 , so the calculated sample size equal 84 patients divided into two equal groups. Included patients were randomized at a 1:1 ratio to "Endoscopic Group, EG" or "Surgical Group , SG" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.(simple random sample). Patients will be divided into 2 groups in accordance type of preoperative

Therapy :

Group 1: "Endoscopic Group, EG" included 42 patients. Group 2: "Surgical Group , SG" included 42 patients.

DETAILED DESCRIPTION:
A- Site of the study: The investigators included all patients who were presented to General Surgery Department with Iatrogenic Esophageal Perforation after Laparoscopic Upper Gastrointestinal Surgery at Zagazig University hospital between (December 2020 to August 2023).

B- Sample size:

The sample size was calculated by using open Epi program depending on the following data ; confidence interval 95% , power of the test 80% , ratio of unexposed/ exposed 1 , the success rate of surgical repair versus endoscopic repair was 98 % versus 75% respectively. Odd ratio 16 , and risk ratio 1.3 , so the calculated sample size equal 84 patients divided into two equal groups.

c- Sample selection: Included patients were randomized at a 1:1 ratio to "Endoscopic Group, EG" or "Surgical Group , SG" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.(simple random sample).

D- Subjects: Patients will be divided into 2 groups in accordance type of preoperative

Therapy :

Group 1: "Endoscopic Group, EG" included 42 patients. Group 2: "Surgical Group , SG" included 42 patients.

Inclusion criteria:

Patients with Iatrogenic Esophageal Perforation after Laparoscopic Upper Gastrointestinal Surgery , failued conservative meaures .patient with good general condition (ASA I&II).

Exclusion criteria:

We excluded patients who bad general condition (ASAIII&IV&V), , respond to conservative measures.

E- Data collection (tools): All patients will subjected to the followings:

patients were selected by randomization method, full history taking, Complete physical examination, laboratory investigations (complete blood picture, liver and kidney functions, coagulation profile, tumor marker tests, serum electrolytes), patients were assessed radio-logically by abdominal &chest x- ray , abdominal ultrasound, pelvic and abdominal CT, upper GI endoscopy.

Study design (operational study):

A. Type of the study : A randomized Controlled Trial.

B. Steps of performance:

1. Complete history taking.
2. Clinical and laboratory results.
3. Radiological results.
4. Endoscopic management of Iatrogenic Esophageal Perforation after Laparoscopic Upper Gastrointestinal Surgery .
5. Analysis of the results.
6. Preparing conclusion and recommendation.

C-Study techniques (procedure):

For patients in EG, we began with assessment of the site & size of perforation . In this study, In this study, we used a fully covered stent (Mega stent, Taewoong Medical Industries, Gyeonggi-do, South Korea) ultra large and long (length: 24 cm, diameter: 36 mm) stent. We did not experience any complication with Mega stent, particularly migration, thanks to the design of Mega stent that fits well for the post-sleeve anatomy with reduction of migration.

Concurrently, the interventional radiology team subcutaneously drained the intraperitoneal free fluid using 2 intra-peritoneal tubes that were placed under US guidance in the sub-hepatic region and in the pelvis.

D-Outcomes:

Primary and secondary outcomes were incidence of postoperative hospital stay and complications in each group during the 3-months follow-up period, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Iatrogenic Esophageal Perforation after Laparoscopic Upper Gastrointestinal Surgery
* failued conservative meaures .
* patient with good general condition (ASA I&II). -

Exclusion Criteria:

* We excluded patients who bad general condition (ASAIII&IV&V),
* respond to conservative measures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
incidence of leak after the intervention | within one week after the procedure
  incidence of leak after the intervention

SECONDARY OUTCOMES:
incidence of side effects of endoscopy | within one month after the surgery
  incidence of side effects of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, MD, Principal Investigator — ZAGAZIG UNIVERSITY HOSPITALS
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: No